CLINICAL TRIAL: NCT03629288
Title: Clinical and Microbiological Efficacy of a Azithromycin as an Adjunct to Non-Surgical Periodontal Treatment : A Randomized Controlled Clinical Trial
Brief Title: Efficacy of Azithromycin as an Adjunct to Non-Surgical Periodontal Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional Andres Bello (Other)
Responsible Party: Principal Investigator, Mariely Navarrete, Associate Professor, Director of Graduate Periodontics Faculty of Dentistry Andres Bello University, Viña del Mar campus, Universidad Nacional Andres Bello
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 038
Record Dates: First submitted 2018-07-02; First posted 2018-08-14 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Periodontitis
Keywords: Azithromycin; Periodontal debridement; Antibiotics; Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Lactose; Azithromycin

STUDY DESIGN:
Intervention Model Description: A double-blind, randomized controlled trial, where patients with a Severe Periodontitis with potencial for additional tooth loss and moderate rate of progression (Stage III grade B). The intervention group received non-surgical periodontal therapy (NSPT) plus azithromycin, and the control group received NSPT plus placebo. The clinical variables were measured before the treatment, and in the first, third and sixth month of the end of the NSPT, while the microbiological variables were measured before the treatment and in the third and sixth month after treatment.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Periodontal treatment, lactose tab (Placebo Comparator): Periodontal treatment (scaling and root planning) and one tablet containing lactose once a day for three days immediately after the scaling and root planning.
  Interventions: Other: Lactose tab
- Periodontal treatment, Antibiotic (Experimental): Periodontal treatment (scaling and root planning) and one tablet containing 500 milligrams (mg) of Azithromycin once a day for three days immediately after the scaling and root planning.
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Other: Lactose tab — Tablet containing lactose Procedure: Periodontal treatment Scaling and root planning
  Arms: Periodontal treatment, lactose tab
Drug: Azithromycin — Tablet containing 500mg Azithromicyn. Procedure: Periodontal treatment Scaling and root planning
  Other Names: Azithromycin 500mg Tab
  Arms: Periodontal treatment, Antibiotic

SUMMARY:
This study evaluates the effect of the systemic administration of azithromycin as a therapy associated with non-surgical periodontal treatment, in the clinical and microbiological variables of patients with Severe Periodontitis with moderate rate of progression (Stage III grade B). A double-blind, randomized, controlled trial was conducted with 18 voluntary patients with a history of moderate to severe chronic periodontitis, who met the inclusion and exclusion criteria and signed an informed consent.

The intervention group received non-surgical periodontal therapy (NSPT) plus azithromycin, and the control group received NSPT plus placebo. Probing Pocket Depth (PPD) Clinical Attachment Level (CAL),O'Leary index (OI) and Bleeding on Probing (BoP) were evaluated as clinical variables while Porphyromonas gingivalis (Pg), Tannerella forsythia (Tf), Treponema denticola (Td), Fusobacterium nucleatum (Fn) were the microbiological variables detected by conventional Polymerase chain reaction (PCR).

DETAILED DESCRIPTION:
Definition of the sample: Patients over 18 years old admitted to the Diagnostic Unit of the Faculty of Dentistry (DUFD), Viña del Mar campus of the Universidad Nacional Andres Bello (UNAB) during 2016, with a diagnosis of severe periodontitis, meeting both the inclusion and exclusion criteria and voluntarily agree to participate of the present research work, signing an informed consent. The chosen participants were informed of the nature of the research, potential risks and compensation for participating in the study, obtaining informed consent from every patient.

Sample Size Calculation: To calculate the minimum sample size necessary for the constitution of the control and intervention groups, the variance of the probing depth difference were considered as fixed values, which were based on the results described above.Considering the above and using a level of significance of 5%, a statistical power of 80% and an estimation error of 1 mm, at least 7 patients were obtained for each group, giving a total of 14 minimum subjects to study.

Protocol and clinical exam: Out of a total of 32 patients who were selected, 20 of those who met the inclusion criteria were randomly assigned by the study coordinator to one of the two groups using a random generation sequence employing a software. Two subjects declined to participate in the research, so the study had 9 participants in each group. In this way, two groups were formed to investigate: an intervention group that received NSPT plus 500 mg of azithromycin once a day for three days immediately after the NSPT, and a control group that received NSPT plus placebo under the same conditions as the intervention group.

Randomization: Only the main investigator, who made the randomization by using the Epidat 4.0 program, had knowledge about the content of the containers and the group to which each patient belonged in the study, therefore, was in charge of labeling the containers, achieving in this way that collaborators and participants in the investigation did not know their content until after the study was finished.

Standardization and calibration: The data was collected using instruments and supplies with the same commercial brands, in a single chair, under the same lighting and by a single examiner in the case of clinical data and another examiner for microbiological variables.

For standardization, measurements were performed under the same conditions and using the same type of instrument, in order to reduce the associated bias. The instruments used for data collection were all the same in design and brand: Basic Examination Kit: Mirror, caries probe, tweezers (Hu-Friedy® Manufacturing Inc., Chicago, IL, USA), manual periodontal probe (North Carolina Probe. Hu-Friedy® Manufacturing Inc., Chicago, IL, USA), plaque finder tablets (Curaprox © CURADEN AG, Switzerland) and number 40 sterile paper cones (Johnson & Johnson, Tokyo, Japan).As there was only one examiner (KL) involved in the study, intra-examiner reliability assessment was executed. This examiner (intra-class correlation coefficient of 0.96 and 0.95 for PPD and CAL), recorded the all stipulated variables, in a clinical file designed especially for the study. Microbiological sampling and NSPT were performed by a single clinician (PO).The complete process of PCR was performed by a biochemist belonging to the microbiology laboratory, Santiago campus of the UNAB.

Periodontopathogens: The presence of periodontopathogens was considered when exposing the agarose gel of the electrophoresis to ultraviolet light, a band at the site of the 197 base pairs (bp) was observed in the lane possessing the patient's subgingival bioflora sample of Pg, 316 base pairs for Td, 745 for Tf and 167 for Fn.

Data collection and instrument: Prior to the data collection, all subjects belonging to the study were asked for a panoramic radiograph for diagnostic purposes. Subsequently, the periodontal examination was performed registering the clinical variables described above in a clinical record.

Obtaining microbiological samples: The microbiological examination was performed before NSPT on both groups. The collection of microbiological samples was based on a protocol that is used at the University of Chile. Using sterile paper cones number 40, a sample of subgingival bioflora was taken from the site with the highest CAL, within those with PD ≥ 5mm, and an oral hygiene instruction was performed. Before the collection of subgingival bioflora, the area was cleaned with a sterile gauze to eliminate the supragingival biofilm. Then, with a tweezer, a paper cone was taken, and its tip was placed in the sulcus of the study site for 20 seconds, to ensure the absorption of the crevicular fluid and subgingival bioflora. Each biological sample obtained was suspended in an Eppendorf tube with 1 ml of distilled water and transported in a refrigerator at a temperature of 4°C approximately, within a time not exceeding 3 hours, to be then temporarily stored at -80°C, until its transfer and subsequent extraction of deoxyribonucleic acid (DNA) and PCR technique processing. The time between sampling and DNA extraction did not exceed 48 hours, to avoid deterioration of the biological material.

Periodontal Treatment: Once the preliminary collection of all the variables was completed, non-surgical periodontal treatment (NSPT) was carried out, beginning with supra and subgingival full-mouth decontamination, using an electric piezo (DTE®, Guilin Woodpecker Medical Instrument Co., Ltd., Guilin, Guangxi , People's Republic of China), followed by root planning at sites presenting PD ≥ 5mm and CAL≥ 4mm, using Gracey curettes (Hu-Friedy® Manufacturing Inc., Chicago, Illinois (IL), USA). This therapy was performed in all patients, both in the intervention and control group, under full mouth treatment protocol, in 1 or 2 work sessions, lasting from 1 to 2 hours, achieving treatment within 24 hours.

Azithromycin or placebo administration: At the end of the last treatment session, the antibiotic azithromycin (Azithromycin, Laboratory Chile) or a placebo (Lactose, Galenic Pharmacy) was administered, depending on the group, intervention or control respectively, to which the patient belonged. For both therapies, the administration regimen was 1 tablet of 500 mg orally per day, for 3 consecutive days.To maintain the double-blind, the containers used for the azithromycin and placebo presented the same characteristics regarding size and color. About the azithromycin tablets and placebo, these were visually identical.

Subsequently, at the first, third and sixth month after the end of the non-surgical treatment, a new collection of all the clinical variables measured at the beginning of the study was performed, while the microbiological variables were measured again at the third and sixth months after treatment, from the same site used in the first sampling.

Statistical Analysis: The analysis of the data was carried out according to the specific objectives of the research, using the Statistical Package for the Social Sciences (SPSS) computer program. A descriptive analysis was performed in which the qualitative variables were studied by frequency, while the quantitative ones were analyzed through the average. The results obtained in both cases were expressed in frequency tables. For each variable, the data normality test was performed according to the Shapiro-Wilk test. Afterwards, an inferential analysis was carried out for the quantitative variables. The level of statistical significance was established according to the Student t and Chi-Square test, while for the qualitative variables, the non-parametric McNemar test was performed. Significant p-values <0.05 were considered, aiming to present a confidence level of 95%.

Ethical implications, biosecurity and others Each patient was informed in detail all that entails carrying out the research work, according to the level of understanding of each subject and was given an informed consent, in which the objective of the study is specified in writing along with the procedures to be performed for both, the control group and the intervention group, in addition to the costs and benefits of participating. The design, together with the protocol of the present study, was based on the Declaration of Helsinki and was approved by the Scientific Ethics Committee of the Faculty of Dentistry, Viña del Mar campus of the UNAB.On the other hand, for the correct development of the investigation, pertinent clinical examinations were carried out following the biosecurity regulations in force at that establishment. The sample taken from the subgingival bioflora of the patient consists of a totally innocuous, fast and simple technique, which was obtained only from a periodontal site. Once the investigation was completed, all the extracted material was destroyed, achieving its elimination by means of the international standards of handling of biological samples. All participants were given free of charge the necessary elements for proper oral hygiene, teaching them the correct way to sanitize their mouth. In addition, they were made aware of the diagnosis, treatment plan and results obtained. Regarding the patients examined who did not meet the inclusion and / or exclusion criteria of the study, they were referred to the subject of Clinical Periodontics for the fourth year, as a teaching assistant or Postgraduate of Periodontics at the UNAB, as appropriate, in order to be treated periodontally. Regarding the use of systemic antibiotics as adjuvant treatment, this has been shown to be clinically more effective than the periodontal treatment associated with placebo. Azithromycin, on the other hand, has an action spectrum that involves aerobic and anaerobic Gram negative bacteria, among which are the periodontopathogens, it has an excellent gastrointestinal absorption, long half-life and limited adverse effects. Due to its properties, it could become a viable alternative in periodontics to the current adjuvant antibiotic regimen of amoxicillin with metronidazole.Regarding the use of the placebo (lactose), it is characterized for being of the pure or inactive type, that is, what corresponds to an inert substance that has no pharmacological action in the patient, which is why it is usually the type of placebo of choice in studies of clinical trials. Lactose is a disaccharide resulting from the binding of glucose and galactose, and these placebos correspond to capsules with a crystalline powder, white, odorless and with a slightly sweet flavor, whose side effects to its use occur infrequently, mainly in patients who have ingested excessive amounts of lactose and / or have intolerance to it, generating symptoms such as abdominal pain, flatulence, diarrhea, bloating, nausea and vomiting.It should be noted that, despite the low prevalence of adverse reactions in both, lactose and azithromycin , patients were warned about the possible effects, indicating that in the face of any discomfort attributable to the consumption of the tablets they would go to the researchers to stop the administration of these and be eliminated from the study.

ELIGIBILITY:
Inclusion criteria:

(I) Patients ≥ 18 years; (II) classified by the American Society of Anesthesiologists (ASA) as ASA I or ASA II that are compatible with local anaesthesia procedures; (III) At least 10 natural teeth present, excluding semi-erupted third molars; (IV) Periodontitis untreated, stage III generalized, grade B, according to the AAP/EFP classification of 2018 29. For Stage III, the following criteria are considered: Severity: Interdental CAL at the site of greatest loss ≥ 5 mm, radiographic bone loss extending to the middle or apical third of the root, and tooth loss due to periodontitis ≤ 4 teeth). Complexity: PPD ≥ 6mm, vertical bone loss ≥ 3mm, furcation involvement Class II or III and Moderate ridge defect. Generalized: >30% of teeth involved. Grade B: Indirect evidence of progression ( % bone loss/age: 0.25 to 1.0)

Exclusion criteria: Patients with (I) Haemostasis disorders; (II) Medication associated with gingival disorders such as: Anticonvulsants (Phenytoin), Calcium channel blockers (Nifedipine), Immunosuppressive drugs (Cyclosporins); (III) Systemic diseases that affect the immunoinflammatory response; (IV) Treatment with antacids on a regular basis due to chronic gastritis and/or self-medication with antacids; (V) Treatment with drugs such as: warfarin, digoxin and acetylsalicylic acid; (VI) History of allergy to local anesthetics; (VII) Orthodontic appliances; (VIII) Antibiotic treatment in the previous 3 months; (IX) History periodontal treatment; (X) Pregnancy; (XI) Valvular prostheses or failures in heart valves, with risk of endocarditis; (XII) Psychic and Intellectual Disability, in accordance with Chilean law number 20,584, title II, paragraph 8, article 28; (XIII) Consumption of more than 10 cigarettes per day; (XIV) Allergy to AZM; (XV) Lactose intolerance.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2016-09-02 (Actual); Study Completion 2016-10-30 (Actual)

PRIMARY OUTCOMES:
Difference between groups (placebo v/s azithromycin) in the mean (±SD) and changes or delta (∆) in number of sites with PPD 1-3 mm, 4-6 mm and ≥ 7 mm in stage III grade B periodontitis patients, before and 1, 3 and 6 months after NSPT. | Baseline,1, 3 and 6 month
  Before, 1, 3 and 6 month after performing NSPT with placebo or azithromycin, PPD was measured in all the patients in the study and corresponds to the distance in millimeters from the gingival margin (MG) to the inserted probe´s tip of the most apical portion of the periodontal pocket. It was obtained by measuring with a North Carolina periodontal probe (Hu-Friedy® Manufacturing Inc., Chicago, IL, USA), from the bottom of the pocket to the MG, in a position parallel to the vertical axis of the tooth, with a pressure no greater than 0.25 Newton (N). PD was performed in a circular direction over the entire surface of each tooth, registering the 6 deepest sites per tooth (mesiobuccal, buccal, distobuccal, distolingual, lingual and mesiolingual).
  Subsequently, those sites with PPD 1-3 mm, 4-6 mm and ≥ 7 mm were counted and the significance of differences between groups at each time point was assessed using the unpaired t-test (p>0.05) or Mann-Whitney U test.

SECONDARY OUTCOMES:
Risk for disease progression, according to Lang & Tonetti (2003). | Baseline and 6 month
  Percentage of subjects presenting low (≤ 4 sites with PPD ≥ 5 mm),moderate (5-8 sites with PPD ≥ 5 mm) or high (≥ 9 sites with PPD ≥5 mm), before and 6 month after performing SRP with placebo or azithromycin.The significance of differences between groups was assessed using the Fisher's exact test (p<0.05).
Clinical Attachment Level (CAL) gain in the sixth month after NSPT with placebo or azithromycin. | Baseline and 6 month
  Before and 6 month after performing NSPT, CAL was measured in all the patients in the study and corresponds to the distance measured in millimeters from the cementum enamel junction to the tip of the probe inserted to the most apical portion of the periodontal pocket. It was obtained using a North Carolina periodontal probe (Hu-Friedy® Manufacturing Inc., Chicago, IL, USA), in a position parallel to the vertical axis of the tooth, with a pressure not greater than 0.25 N.
Difference between groups for the O'Leary index (OI),in stage III grade B periodontitis patients before and 1, 3 and 6 month after performing NSPT with placebo or azithromycin. | Baseline,1, 3 and 6 month
  Before,1,3 and 6 month after performing NSPT, OI was measured in all the patients in the study. OI is percentage of dental surfaces with staining, through the use of biofilm developers. To obtain the index, a curaprox developer tablet was dissolved in a plastic cup with water and with a cotton ball this solution was applied on all of the tooth surfaces, recording only those that were stained. The calculation was made by dividing the surfaces that stained by the total surfaces, which corresponds to the number of teeth present multiplied by 4, and multiplying this value by 100. Subsequently, the significance of differences between groups at each time point was assessed using the unpaired t-test and x2 test (p<0.05)
Difference between groups for the bleeding on probing (BoP) Index, in stage III grade B periodontitis patients before and 1, 3 and 6 month after performing NSPT with placebo or azithromycin. | Baseline,1, 3 and 6 month
  Before,1, 3 and 6 month after performing NSPT, BoP was measured in all the patients in the study. BoP is the percentage of surfaces that bleed when probing. It was recorded during PPD measurement with a North Carolina periodontal probe (Hu-Friedy® Manufacturing Inc., Chicago, IL, USA) and was considered positive if it occurs 30 seconds after probing. The calculation was made by dividing the sites that bled by the total sites, which corresponds to the number of teeth present multiplied by 6, and multiplying this value by 100. Subsequently, the significance of differences between groups at each time point was assessed using the unpaired t-test and x2 test (p<0.05)
Presence of periodontopathogens before, 3 and 6 month after performing NSPT with placebo or azithromycin. | Baseline, 3 and 6 month
  Before, 3 and 6 month after performing NSPT, the microbiological examination was performed on both groups. The biofilm samples were analyzed to detect the presence of four bacterial species: Porphyromonas gingivalis (Pg), Tannerella forsythia (Tf), Treponema denticola (Td), Fusobacterium nucleatum (Fn) by Polymerase chain reaction (PCR).Subsequently,the significance of differences between groups at each time point was assessed using the unpaired t-test and x2 test (p<0.05)

CONTACTS AND LOCATIONS:
Overall Officials: Mariely A Navarrete, MSc, Study Director — Universidad Nacional Andres Bello; Mariely A Navarrete, MSc, Principal Investigator — Universidad Nacional Andres Bello
Locations (1):
- Universidad Nacional Andres Bello, Viña del Mar, Región de Valparaíso, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tonetti MS, Greenwell H, Kornman KS. Staging and grading of periodontitis: Framework and proposal of a new classification and case definition. J Periodontol. 2018 Jun;89 Suppl 1:S159-S172. doi: 10.1002/JPER.18-0006. PMID 29926952
- [Background] Meissner K, Bingel U, Colloca L, Wager TD, Watson A, Flaten MA. The placebo effect: advances from different methodological approaches. J Neurosci. 2011 Nov 9;31(45):16117-24. doi: 10.1523/JNEUROSCI.4099-11.2011. PMID 22072664
- [Background] Suchy FJ, Brannon PM, Carpenter TO, Fernandez JR, Gilsanz V, Gould JB, Hall K, Hui SL, Lupton J, Mennella J, Miller NJ, Osganian SK, Sellmeyer DE, Wolf MA. National Institutes of Health Consensus Development Conference: lactose intolerance and health. Ann Intern Med. 2010 Jun 15;152(12):792-6. doi: 10.7326/0003-4819-152-12-201006150-00248. Epub 2010 Apr 19. No abstract available. PMID 20404261
- [Background] Jellema P, Schellevis FG, van der Windt DA, Kneepkens CM, van der Horst HE. Lactose malabsorption and intolerance: a systematic review on the diagnostic value of gastrointestinal symptoms and self-reported milk intolerance. QJM. 2010 Aug;103(8):555-72. doi: 10.1093/qjmed/hcq082. Epub 2010 Jun 3. PMID 20522486
- [Result] Sampaio E, Rocha M, Figueiredo LC, Faveri M, Duarte PM, Gomes Lira EA, Feres M. Clinical and microbiological effects of azithromycin in the treatment of generalized chronic periodontitis: a randomized placebo-controlled clinical trial. J Clin Periodontol. 2011 Sep;38(9):838-46. doi: 10.1111/j.1600-051X.2011.01766.x. Epub 2011 Jul 19. PMID 21770996
- [Result] Lang NP, Tonetti MS. Periodontal risk assessment (PRA) for patients in supportive periodontal therapy (SPT). Oral Health Prev Dent. 2003;1(1):7-16. PMID 15643744